CLINICAL TRIAL: NCT05661357
Title: Single Arm, Prospective, Exploratory Clinical Study of Disitamab Vedotin Combined With Fruquintinib for Advanced Colorectal Cancer With HER2 Expression or Mutation That Has Received at Least Two Standard Treatment Failures
Brief Title: Disitamab Vedotin Combined With Fruquintinib for mCRC With HER2 Expression
Acronym: HCCSC-C03
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Collaborators: Huangshi Central Hospital (Other); The First People's Hospital of Tianmen (Unknown); Sir Run Run Shaw Hospital (Other); Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, Prof, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC C03
Record Dates: First submitted 2022-11-08; First posted 2022-12-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: HER2; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin combined with Fruquintinib (Experimental): Single arm, prospective, exploratory clinical study of Disitamab Vedotin combined with Fruquintinib for advanced colorectal cancer with HER2 expression or mutation that has received at least two standard treatment failures
  Interventions: Drug: Disitamab Vedotin Combined With Fruquintinib

INTERVENTIONS:
Drug: Disitamab Vedotin Combined With Fruquintinib — Furquinotinib: 3mg, Qd, 28 days as a cycle. Vidicizumab: according to the instructions of Vidicizumab, d1, 2.5 mg/kg, intravenous drip (ivgtt)

SUMMARY:
Single arm, prospective, exploratory clinical study of Disitamab Vedotin combined with Fruquintinib for advanced colorectal cancer with HER2 expression or mutation that has received at least two standard treatment failures

DETAILED DESCRIPTION:
Colorectal cancer is the fourth deadliest malignant tumor in the world, and the 5-year survival rate of patients with advanced colorectal cancer is only 12%. In September 2018, furoquentinib was the first approved in China for the treatment of metastatic colorectal cancer patients who failed to receive at least two systematic anti-tumor treatments. The FRESCO trial is a multicenter (28 hospitals in China), randomized, double-blind and placebo controlled phase III trial, The median OS of patients receiving furoxigenib was 9.3 months, while the mOS of patients receiving placebo was 6.57 months (HR=0.65, 95% CI: 0.51~0.83, P<0.001); As a secondary endpoint, mPFS was 3.71 and 1.84 months (HR=0.26, 95% CI: 0.21~0.34, P<0.001). In order to further improve the efficacy, it is necessary to continue to explore the combined treatment strategy of furoquentinib: combined chemotherapy, other targeted treatment and local treatment may benefit more CRC patients. HER2 amplification or overexpression was found in 2%~6% of patients with advanced or metastatic colorectal cancer. In the past decade, several studies have identified it as a potential target for the treatment of HER2 positive colorectal cancer, and it has been written into the guidelines for posterior line therapy. The prognostic value of HER2 overexpression in advanced colorectal cancer is still unclear. The anti-tumor activity of dual targeted HER2 treatment schemes, such as Patuzumab+Trastuzumab, Trastuzumab+Tucatinib, Trastuzumab+Lapatinib, has been significantly increased, which has been confirmed in clinical studies. Vidiximab contains a new humanized anti HER2 antibody Disitamab, which is coupled to monomethylolestatin E (MMAE) through a cleavable linker. Its antibody has a high affinity for HER2 and can efficiently bind with it and enter cancer cells; The linker is cleavable in the tumor cell membrane, which can rapidly release small molecule cytotoxic drugs, and has a bystander killing effect against heterogeneous tumor cells. This one arm, prospective, open study was designed to explore the efficacy and safety of vidiximab combined with furoquentinib triple line or above in the treatment of advanced colorectal cancer with HER2 expression or mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer patients aged ≥ 18 years and ≤ 75 years;
2. ECOG score 0-1;
3. Patients with advanced colorectal cancer who are pathologically diagnosed as HER2 expression or mutation and who fail or are intolerant after second-line treatment; Note: HER2 expression refers to patients with tumor cell immunohistochemical staining intensity of 1+, 2+or 3+confirmed to have expression at least once in the pathological detection/review of primary or metastatic lesions conducted by the pathology department of our hospital, or patients with advanced colorectal cancer with HER2 gene amplification or mutation confirmed by NGS.
4. According to RECIST 1.1 standard, there is at least one measurable target lesion, and tumor imaging evaluation is conducted within 28 days before the first drug use;
5. Estimated survival time ≥ 12 weeks;
6. If the main organs function normally, they meet the following standards:

(1) The blood routine examination standard should meet: ANC ≥ 1.5 × 109/L； PLT ≥90 × 109/L； Hb ≥ 90g/L (no blood transfusion within 14 days); (2) Biochemical examination shall meet the following standards: ALB ≥ 30g/L; (No ALB within 14 days); TBIL ≤ upper limit of normal value (ULN); ALT and AST ≤ 2.5 times the upper limit of normal value (ULN). If there is liver metastasis, ALT and AST ≤ 5ULN; Alkaline phosphatase ≤ 2.5 times the upper limit of normal value (ULN); BUN and Cr ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min (Cockcroft Gault formula); (3) Color Doppler echocardiography and echocardiography: left ventricular ejection fraction (LVEF ≥ 50%); (4) QT interval (QTcF) corrected by Fridericia method of 12 lead ECG in women<470 ms; 7. For female patients without menopause or surgical sterilization: during the treatment period and at least 7 months after the last administration of the drug in the study treatment, agree to abstinence or use effective contraception methods; 8. Volunteer to join the study and sign the informed consent form.

Exclusion Criteria:

1. Have received anti-tumor treatment or radiotherapy for any malignant tumor in the past;
2. At the same time, they received anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphate therapy or immunotherapy;
3. The patient has undergone major surgery unrelated to colorectal cancer within 4 weeks before enrollment, or the patient has not fully recovered from such surgery;
4. Serious heart disease or discomfort, including but not limited to the following diseases:

   * History of diagnosis of heart failure or systolic dysfunction (LVEF<50%)
   * High risk uncontrolled arrhythmia, such as atrial tachycardia, resting heart rate>100 bpm, significant ventricular arrhythmia (such as ventricular tachycardia) or higher grade atrioventricular block (i.e. Mobitz II second degree atrioventricular block or third degree atrioventricular block)
   * Angina requiring anti angina drugs
   * Valvular heart disease with clinical significance
   * ECG showed transmural myocardial infarction
   * Poor control of hypertension (systolic blood pressure>180 mmHg and/or diastolic blood pressure>100 mmHg)
5. Inability to swallow, intestinal obstruction or other factors affecting drug administration and absorption;
6. People known to have a history of allergy to the drug components of this protocol; Have a history of immunodeficiency, including HIV test positive, HBV/HCV test positive, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
7. Women in pregnancy and lactation, women with fertility and positive baseline pregnancy test, or women in childbearing age who are unwilling to take effective contraceptive measures during the whole trial period and within 7 months after the last study drug use;
8. Suffer from serious concomitant diseases or other concomitant diseases that may interfere with the planned treatment, or The investigator believes that the patient is not suitable to participate in any other situation of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, an average of 2 years
  Objective Response Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No